CLINICAL TRIAL: NCT01385189
Title: Phase I Study of the Safety and Immunogenicity of Na-GST-1/Alhydrogel® With Different Doses of the Novel Immunostimulant GLA-AF in Healthy Adults
Brief Title: Safety and Immunogenicity of a Human Hookworm Candidate Vaccine With Different Doses of a Novel Adjuvant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Children's National Research Institute (Other); George Washington University (Other)
Responsible Party: Principal Investigator, Maria Elena Bottazzi PhD, Sponsor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SVI-11-01
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Hookworm Infection; Hookworm Disease
Keywords: Human Hookworm Vaccine Initiative; HHVI; Human Hookworm; Hookworm; Hookworm Disease; N. americanus; Soil-transmitted helminth infection; Intestinal blood loss; Iron deficiency anemia
MeSH Terms: conditions — Hookworm Infections; Ancylostomiasis; Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental): 10 μg Na-GST-1/Alhydrogel vs. 10 μg Na-GST-1/Alhydrogel/GLA-AF (1 μg)
  Interventions: Biological: 10 μg Na-GST-1/Alhydrogel; Biological: 10 μg Na-GST-1/Alhydrogel/GLA-AF (1 μg)
- Cohort 2 (Experimental): 30 μg Na-GST-1/Alhydrogel vs. 30 μg Na-GST-1/Alhydrogel/GLA-AF (1 μg)
  Interventions: Biological: 30 μg Na-GST-1/Alhydrogel; Biological: 30 μg Na-GST-1/Alhydrogel/GLA-AF (1 μg)
- Cohort 3 (Experimental): 30 μg Na-GST-1/Alhydrogel/GLA-AF (5 μg)
  Interventions: Biological: 30 μg Na-GST-1/Alhydrogel/GLA-AF (5 μg)
- Cohort 4 (Experimental): 100 μg Na-GST-1/Alhydrogel/GLA-AF (1 μg)
  Interventions: Biological: 100 μg Na-GST-1/Alhydrogel
- Cohort 5 (Experimental): 100 μg Na-GST-1/Alhydrogel/GLA-AF (5 μg)
  Interventions: Biological: 100 μg Na-GST-1/Alhydrogel/GLA-AF (5 μg)

INTERVENTIONS:
Biological: 10 μg Na-GST-1/Alhydrogel — 3 doses 10 μg Na-GST-1/Alhydrogel administered at 56 day intervals
  Arms: Cohort 1
Biological: 30 μg Na-GST-1/Alhydrogel — 3 doses 30 μg Na-GST-1/Alhydrogel administered at 56 day intervals
  Arms: Cohort 2
Biological: 100 μg Na-GST-1/Alhydrogel — 3 doses 100 μg Na-GST-1/Alhydrogel administered at 56 day intervals
  Arms: Cohort 4
Biological: 10 μg Na-GST-1/Alhydrogel/GLA-AF (1 μg) — 3 doses 10 μg Na-GST-1/Alhydrogel/GLA-AF (1 μg) administered at 56 day intervals
  Arms: Cohort 1
Biological: 30 μg Na-GST-1/Alhydrogel/GLA-AF (1 μg) — 3 doses of 30 μg Na-GST-1/Alhydrogel/GLA-AF (1 μg) administered at 56 day intervals
  Arms: Cohort 2
Biological: 30 μg Na-GST-1/Alhydrogel/GLA-AF (5 μg) — 3 doses 30 μg Na-GST-1/Alhydrogel/GLA-AF (5 μg) administered at 56 day intervals
  Arms: Cohort 3
Biological: 100 μg Na-GST-1/Alhydrogel/GLA-AF (5 μg) — 3 doses 100 μg Na-GST-1/Alhydrogel/GLA-AF (5 μg) administered at 56 day intervals
  Arms: Cohort 5

SUMMARY:
This study is designed to evaluate the safety, reactogenicity, and immunogenicity of Na-GST-1 adsorbed to Alhydrogel® with or without two different dose concentrations of a novel adjuvant, GLA-AF (1 µg or 5 μg) among healthy adult volunteers.

DETAILED DESCRIPTION:
Human hookworm infection is a soil-transmitted helminth infection caused by the nematode parasites Necator americanus and Ancylostoma duodenale. It is one of the most common chronic infections of humans, afflicting up to 740 million people in the developing nations of the tropics. The largest number of cases occurs in impoverished rural areas of sub-Saharan Africa, Southeast Asia, China, and the tropical regions of the Americas. Approximately 3.2 billion people are at risk for hookworm infection in these areas. N. americanus is the most common hookworm worldwide, whereas A. duodenale is more geographically restricted.

The primary approach to hookworm control worldwide has been the frequent and periodic mass administration of benzimidazole anthelminthics to school-aged children living in high-prevalence areas. In 2001, the World Health Assembly adopted Resolution 54.19 which urges member states to provide regular anthelminthic treatment to high-risk groups with the target of regular treatment of at least 75% of all at-risk school-aged children. However, the cure rates for a single dose of a benzimidazole varies with rates as low as 61% (400 mg) and 67% (800 mg) for albendazole and 19% (single dose) and 45% (repeated dose) for mebendazole being reported. These concerns have prompted interest in developing alternative tools for hookworm control. Vaccination to prevent the anemia associated with moderate and heavy intensity hookworm infection would alleviate the public health deficiencies of drug treatment alone.

The current strategy for development of Human Hookworm candidate vaccines is focused on antigens expressed during the adult stage of the hookworm life cycle which play a role in digesting the host hemoglobin, used by the worm as an energy source. These antigens are relatively hidden from the human immune system during natural infection, and hence have a low likelihood of inducing antigen-specific IgE in exposed/infected individuals, reducing the potential for allergic reaction upon vaccination.

The nutritional and metabolic requirements of the adult hookworm living in the human intestine are dependent upon degradation of host hemoglobin that has been ingested by the worm. N. americanus hookworms depend on host hemoglobin for survival. Following hemolysis, adult hookworms use an ordered cascade of hemoglobinases to cleave hemoglobin into smaller molecules. Following hemoglobin digestion, the freed heme generates toxic oxygen radicals that can be bound and detoxified by molecules such as glutathione S-transferase-1 (GST-1). GST-1 of N. americanus (Na-GST-1) is a critical enzyme that plays a role in parasite blood feeding; when used as a vaccine, the investigators hypothesize that the antigen will induce anti-enzyme neutralizing antibodies that will interfere with parasite blood-feeding and cause parasite death or reduce worm fecundity.

Following its selection as a candidate antigen Na-GST-1 has been successfully manufactured and tested in the laboratory and in animals with both Alhydrogel® (aluminum hydroxide suspension)and Alhydrogel® plus Gluco-Pyranosylphospho-Lipid A Aqueous Formulation (GLA-AF). Na-GST-1 has been shown to be pure, potent, and stable when administered as either of these two formulations.

Although GLA-AF has not yet been administered to humans, an oil-in-water emulsion of GLA (GLA-SE) has been used in combination with the Fluzone® trivalent killed influenza vaccine in a Phase 1 trial. In this study, doses up to 1 µg of GLA-SE were safe and well-tolerated and significantly enhanced influenza-specific antibody responses.

The phase 1 trial described here will enroll healthy adults who have not been infected with or exposed to hookworm who are living in the Washington DC area. A phase 1 trial of Na-GST-1/Alhydrogel (with or without GLA-AF) is planned to start in July 2011 in Brazil. In that study, both hookworm-naïve and hookworm-exposed healthy adults will be vaccinated with either Na-GST-1/Alhydrogel®, Na-GST-1/Alhydrogel® co-administered with 1 µg GLA-AF, or the Butang® hepatitis B vaccine. The objectives of that study will be to assess the safety and immunogenicity of the Na-GST-1 formulations in healthy Brazilian adults. The study described here will complement the study in Brazilian adults as it will provide additional information about different dose concentrations of GLA-AF as well as detailed data on the humoral immune response to the different formulations that will be tested.

In this study, 90 volunteers will be progressively enrolled into one of six dose cohorts. Dose cohorts will be enrolled and vaccinated in a consecutive fashion. The 15 volunteers in each cohort will be subsequently randomized in a 1:2 ratio to receive either the Na-GST-1/Alhydrogel® (n=5) or Na-GST-1/Alhydrogel®/GLA-AF (n=10). In the first, third and fifth cohorts, volunteers will be randomized to receive either Na-GST-1/Alhydrogel® (n=5) OR Na-GST-1/Alhydrogel® co-administered with 1 µg GLA-AF (n=10), while in the second, fourth, and sixth cohorts, volunteers will be randomized to receive either Na-GST-1/Alhydrogel® (n=5) or Na-GST-1/Alhydrogel® co-administered with 5 µg GLA-AF (n=10).

Each participant will receive 3 doses of the assigned study agent given in 56 day intervals (i.e. Day 0, Day 56 and Day 112). The trial is expected to last for approximately 18 months. Each participant will be followed for 16 months from the time of the first injection.

Safety parameters will be monitored throughout the study. The primary endpoint for the study will be measurement of antigen-specific antibody response.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 45 years, inclusive.
* Good general health as determined by means of the screening procedure.
* Available for the duration of the trial (16 months).
* Willingness to participate in the study as evidenced by signing the informed consent document.

Exclusion Criteria:

* Pregnancy as determined by a positive urine β-hCG (if female).
* Participant unwilling to use reliable contraception methods up until one month following the third immunization (if female).
* Currently lactating and breast-feeding (if female).
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, diabetes, or renal disease by history, physical examination, and/or laboratory studies.
* Known or suspected immunodeficiency.
* Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25-times the upper reference limit).
* Laboratory evidence of renal disease (serum creatinine greater than 1.25-times the upper reference limit, or more than trace protein or blood on urine dipstick testing).
* Laboratory evidence of hematologic disease (hemoglobin <12.5 g/dl [females] or <13.5 g/dl [males]; absolute leukocyte count <3500/mm-cubed or >10.5 x 103/mm-cubed; absolute neutrophil count [ANC] <2000/ mm-cubed; absolute lymphocyte count <1100/mm-cubed; or platelet count <140,000/mm-cubed).
* Laboratory evidence of a coagulopathy (PTT or PT INR greater than 1.1-times the upper reference limit).
* Serum glucose (random) greater than 1.2-times the upper reference limit.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
* Participation in another investigational vaccine or drug trial within 30 days of starting this study.
* Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma as defined by the need for regular use of inhalers or emergency clinic visit or hospitalization within the last 6 months.
* Positive ELISA for HBsAg.
* Positive ELISA and confirmatory Western blot tests for HIV-1.
* Positive ELISA and confirmatory immunoblot tests for HCV.
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study.
* Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to entry into the study.
* History of a surgical splenectomy.
* Receipt of blood products within the past 6 months.
* History of allergy to yeast.
* History of previous infection with hookworm or residence for more than 6 months in a hookworm-endemic area.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Diemert, MD, Study Director — Albert B. Sabin Vaccine Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Diemert DJ, Freire J, Valente V, Fraga CG, Talles F, Grahek S, Campbell D, Jariwala A, Periago MV, Enk M, Gazzinelli MF, Bottazzi ME, Hamilton R, Brelsford J, Yakovleva A, Li G, Peng J, Correa-Oliveira R, Hotez P, Bethony J. Safety and immunogenicity of the Na-GST-1 hookworm vaccine in Brazilian and American adults. PLoS Negl Trop Dis. 2017 May 2;11(5):e0005574. doi: 10.1371/journal.pntd.0005574. eCollection 2017 May. PMID 28464026
- Available data/document: Clinical Study Report — http://smhs.gwu.edu/mitm-crg/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 12 | 12 | 4 | 4 | 8
Completed | 11 | 11 | 4 | 3 | 6
Not Completed | 1 | 1 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 12 | 12 | 4 | 4 | 8 | 40
Age, Continuous [Mean (Full Range); unit: years] | 34.3 [18 to 45] | 33.8 [18 to 45] | 26.3 [18 to 33] | 23.3 [18 to 39] | 35.0 [26 to 45] | 32.9 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 1 | 1 | 5 | 16
  Male | 8 | 7 | 3 | 3 | 3 | 24

OUTCOME MEASURES:

1. Primary Outcome: Immediate Vaccine Related Adverse Events
Description: Frequency of vaccine-related AEs, graded by severity, for each dose and formulation of Na-GST-1
Time Frame: 2 hours post vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 12 | 12 | 4 | 4 | 8
Participants | 4 | 1 | 0 | 1 | 4

2. Secondary Outcome: IgG Antibody Response to Na-GST-1
Description: Dose and formulation of Na-GST-1 that generates the highest IgG antibody response at Day 126, as determined by an indirect enzyme-linked immunosorbent assay (ELISA)
Time Frame: 126 days post dose 1
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | 10 μg Na-GST-1/Alhydrogel | 10 µg Na-GST-1/Alhydrogel/GLA-AF (1 µg) | 30 µg Na-GST-1/Alhydrogel | 30 µg Na-GST-1/Alhydrogel/GLA-AF (1 µg) | 30 µg Na-GST-1/Alhydrogel/GLA-AF (5 µg) | 100 µg Na-GST-1/Alhydrogel | 100 µg Na-GST-1/Alhydrogel/GLA-AF (5 µg)
Number analyzed (Participants) | 4 | 7 | 3 | 7 | 4 | 3 | 6
Arbitrary Units | 17.12 (24.11) | 210.02 (366.67) | 66.86 (105.60) | 64.65 (74.86) | 69.34 (107.46) | 117.24 (117.99) | 89.42 (97.80)

ADVERSE EVENTS:
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/4 | 0/4 | 1/8
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12 | 4/4 | 4/4 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=12) | Cohort 2 (N=12) | Cohort 3 (N=4) | Cohort 4 (N=4) | Cohort 5 (N=8)
Delusional Episode (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study intervention. Full recovery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=12) | Cohort 2 (N=12) | Cohort 3 (N=4) | Cohort 4 (N=4) | Cohort 5 (N=8)
Injection Site Pain (General disorders) | 6 (13) | 4 (8) | 3 (5) | 1 (3) | 5 (8)
Injection Site Tenderness (General disorders) | 4 (9) | 5 (9) | 3 (6) | 2 (2) | 4 (8)
Injection Site Erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection Site Swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 8 (11) | 7 (10) | 2 (4) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthrlagia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No